CLINICAL TRIAL: NCT01660789
Title: "Fit For Kids" Copenhagen - an Interventions Study on Obesity and Physical Inactivity in Children.
Brief Title: "Fit For Kids"-Copenhagen
Acronym: FFK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Inge Holm, Administrator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2-2011-132
Record Dates: First submitted 2012-04-02; First posted 2012-08-09 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Obesity
Keywords: Obesity; Diabetes; Physical activity
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Motor Activity | interventions — Exercise; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle intervention (Other): Lifestyle intervention.
  Interventions: Behavioral: Physical activity, dietary counseling, coaching

INTERVENTIONS:
Behavioral: Physical activity, dietary counseling, coaching — Physical activity, dietary counseling, coaching

SUMMARY:
This study aims to evaluate the effect of a 40- week multifactorial intervention against overweight, obesity and physical inactivity in Danish children.

The investigators wish to examine 40 children before and after the "Fit for Kids" intervention with basic anthropometric measures such as body mass indexi (BMI), waist/hip ratio, systolic- and diastolic blood pressure, level of physical fitness and Total Body fat mass.

Furthermore the investigators wish to examine the more specific inflammatory, metabolic and hormonal effect of the intervention with a more extensive examination programme.

The tests include a DXA-scan, cardio-respiratory fitness, accelerometer monitoring, pedometer monitoring, cognitive testing, Continuous Glucose Monitoring System, different metabolic and inflammatory markers and an oral glucose tolerance test. The study will take place at Centre of Inflammation and Metabolism, Rigshospitalet, Copenhagen.

The study is a randomised controlled trial with a gradual rollout. The 40 children will be randomised. Twenty children will start the intervention at baseline and 20 children will start after the first 20 weeks of intervention, thus providing a control group.

The investigators expect to find a significant reduction in BMI, total body fat mass and systolic blood pressure after the intervention. As for the more extensive tests, the data approach is explorative, as the investigators look at more statistical dependent variables. The contribution of this project is a further description on the effect of intervention against overweight and physical inactivity on the metabolic and inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* Obese children

Exclusion Criteria:

* Other chronic medical conditions
* Medical intake

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
BMI | One year

CONTACTS AND LOCATIONS:
Overall Officials: Nina Marie Birk Eriksen, MD, Principal Investigator — Centre of Inflammation and Metabolism
Locations (1):
- Centre of Inflammation and Metabolism, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Harder-Lauridsen NM, Birk NM, Ried-Larsen M, Juul A, Andersen LB, Pedersen BK, Krogh-Madsen R. A randomized controlled trial on a multicomponent intervention for overweight school-aged children - Copenhagen, Denmark. BMC Pediatr. 2014 Oct 21;14:273. doi: 10.1186/1471-2431-14-273. PMID 25330848